CLINICAL TRIAL: NCT01145339
Title: A Phase III, Non-Inferiority, Randomized, Double-Blind, Parallel-Group, Multicentre, Single-Dose, Comparative Clinical Study of Lactase Eurofarma (Test Drug) and Lactaid® (Comparative Drug), Assessing the Efficacy and Safety in the Treatment of Patients With Lactose Intolerance (Hypolactasia)
Brief Title: A Non-inferiority, Multicenter and Randomized, Single-Dose Study About a Treatment to Hypolactasia (LAILAI)
Acronym: EF099
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EF099
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2011-10

CONDITIONS: Hypolactasia
MeSH Terms: conditions — Lactose Intolerance | interventions — Lactase

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactase EUF (Experimental): 1 chewable tablet of the test drug 30 minutes before the standard lactose dose (25 g).
  Interventions: Drug: Lactase
- Lactase Ref (Active Comparator): 1 chewable tablet of the comparative drug 30 minutes before the standard lactose dose (25 g).
  Interventions: Drug: Lactase

INTERVENTIONS:
Drug: Lactase — 1 chewable tablet of the test drug or comparative drug 30 minutes before the standard lactose dose (25 g).

SUMMARY:
The study primary objective is to compare the clinical efficacy of two formulations in the supportive treatment of lactose intolerance.

ELIGIBILITY:
Inclusion Criteria:

1. The patient should be a male or female, aged between 18 and 60 years old;
2. Have a medical history consistent with lactose intolerance, confirmed by the test of hydrogen in the expired air;
3. The female patients should agree to use birth control methods during the study participation;
4. To be able to meet the study instructions and all the visits required;
5. To give a free consent to participate in the study and sign the informed consent form (ICF).

Exclusion Criteria:

1. Smoking;
2. Secondary hypolactasia;
3. Gastrointestinal inflammatories diseases - present diverticular disease, diabetic gastropathy or neoplasias;
4. Colonoscopy or colon cleaning procedure 4 weeks before the start of study
5. Latrogenic: unnoticed intake of laxatives in over-the-counter drugs or alternative medicine, intake of cereal bran or probiotics;
6. Diagnosis of HIV, immunodepression of any origin, or cancer under treatment.
7. Diagnosis of other comorbidity that, at the investigator's discretion, may compromise the study participation (e.g., systemic infection during the study or use of antibiotics in the last 4 weeks, diabetes mellitus, uncontrolled hypertension or renal failure),
8. Hypersensitivity or previous laboratory or clinical adverse event related to the use of lactase or any of the components of the formulations used in the study;
9. Incapacity to understand and complete the study questionnaires, including the questions that require the use of the Visual Analogue Scale and ICF;
10. Pregnancy or lactation;
11. Use of alcohol, exceeding 3 doses daily;
12. Participation in another clinical study on the last 12 months;
13. Patient having some chronic pulmonary disease that, in the investigator's opinion, may harm or interfere with the expired hydrogen test (e.g., cystic fibrosis).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2011-07; Primary Completion 2011-11 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Hydrogen value in the air expired | 03 times
  Hydrogen value in the expired air for 3h after the patient exposure to the standardized Lactose 25g dose with interventional exogenous Lactase (comparative and test drugs).

CONTACTS AND LOCATIONS:
Overall Officials: Aderson Damião, M.D, Principal Investigator — Hospital das Clínicas de São Paulo; Heda Amarante, M.D, Principal Investigator — Hospital Nossa Senhora das Graças; Marta Machado, M.D, Principal Investigator — Hospital São Lucas PUCRS; Sender Miszputen, M.D, Principal Investigator — Hospital São Paulo / UNIFESP; Wilson Catapani, M.D, Principal Investigator — Faculdade de Medicina do ABC; Mauro Bafutto, M.D, Principal Investigator — Instituto Goiano de Gastroenterologia; Carlos Francesconi, M.D, Principal Investigator — Hospital Mãe de Deus; Maria do Carmo Passos, M.D, Principal Investigator — Instituto Alfa de Gastroenterologia de BH
Locations (7):
- Brazil (7):
  - Instituto Goiano de Gastroenterologia, Goiânia, Goiás
  - Instituto Alfa de Gastroenterologia, Belo Horizonte, Minas Gerais
  - Hospital Nossa Senhora das Graças, Curitiba, Paraná
  - Hospital São Lucas, Porto Alegre, Rio Grande do Sul
  - Hospital Mãe de Deus, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Hospital São Paulo / UNIFESP, São Paulo, São Paulo